CLINICAL TRIAL: NCT03994484
Title: Pharmacokinetics of Single and Multiple Doses of HA121-28 Tablets and Exploration of Maximum Tolerated Dose in Patients With Advanced Solid Tumor in PhaseⅠClinical Trial
Brief Title: Study of Dosage Exploration and Pharmacokinetics for HA121-28 Tablets
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HA121-28/2017/01
Record Dates: First submitted 2019-06-18; First posted 2019-06-21 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HA121-28 tables (Experimental): Participants will receive oral HA121-28 at a starting dose of 25 mg once daily at the 1st day in 0 cycle and for 21 days on a 28-day treatment cycle
  Interventions: Drug: HA121-28 tablets

INTERVENTIONS:
Drug: HA121-28 tablets — Participants will receive oral HA121-28 at a starting dose of 25 mg once daily at the 1st day in 0 cycle and for 21 days on a 28-day treatment cycle
Drug: HA121-28 tablets — Participants will receive oral HA121-28 at a dose of 50 mg once daily at the 1st day in 0 cycle and for 21 days on a 28-day treatment cycle
Drug: HA121-28 tablets — Participants will receive oral HA121-28 at a dose of 100 mg once daily at the 1st day in 0 cycle and for 21 days on a 28-day treatment cycle
Drug: HA121-28 tablets — Participants will receive oral HA121-28 at a dose of 200 mg once daily at the 1st day in 0 cycle and for 21 days on a 28-day treatment cycle
Drug: HA121-28 tablets — Participants will receive oral HA121-28 at a dose of 300 mg once daily at the 1st day in 0 cycle and for 21 days on a 28-day treatment cycle
Drug: HA121-28 tablets — Participants will receive oral HA121-28 at a dose of 450 mg once daily at the 1st day in 0 cycle and for 21 days on a 28-day treatment cycle
Drug: HA121-28 tablets — Participants will receive oral HA121-28 at a dose of 600 mg once daily at the 1st day in 0 cycle and for 21 days on a 28-day treatment cycle
Drug: HA121-28 tablets — Participants will receive oral HA121-28 at a dose of 800 mg once daily at the 1st day in 0 cycle and for 21 days on a 28-day treatment cycle

SUMMARY:
There are 2 phases in this study: Phase 1 (dose escalation) and Phase 2 (dose expansion).

The goal of Phase 1 of this clinical research study is to find the highest tolerable dose of HA121-28 tablets that can be given to patients with advanced cancer. The goal of Phase 2 of this study is to learn if the dose of HA121-28 tablets found in Phase 1 can help to control advanced cancer.

The safety of HA121-28 tablets will be studied in both phases of the study.

DETAILED DESCRIPTION:
If participants are found to be eligible to take part in this study, they will be assigned to a study group based on when they join this study. Up to 8 groups of up to 20 participants will be enrolled in Phase 1 of the study, and up to 3 groups of up to 24 participants will be enrolled in Phase 2.

If participant is enrolled in Phase 1, the dose of HA121-28 tablets they receive will depend on when they join this study. The first group of participants will receive the lowest dose level of HA121-28 tablets. Each new group will receive a higher dose of HA121-28 tablets than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of HA121-28 tablets is found. If participant is enrolled in Phase 2, they will receive HA121-28 tablets at the low, medium and high doses to select the recommended dose for phase Ⅱ clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing to participate in the clinical trial and sign the informed consent;
2. Men and women aged 18 to 75 years;
3. Histologically/cytologically confirmed advanced/metastatic solid tumor, and have failed prior standard therapy or for which no standard therapy is durable(patients with RET fusion/mutation can be included regardless of whether they have received standard therapy or not);
4. At least one measurable lesion according to RECIST 1.1 ;
5. Subject has not received any anti-cancer therapies including chemotherapy, radiotherapy, targeted treatment and surgery within 4 weeks prior to participation;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0~1;
7. Expected overall survival (Life expectancy)≥ 3 months;
8. Laboratory test results must meet the following standards:

   Absolute neutrophil count (ANC) ≥1.5 x 10^9/L; Platelet count (PLT) ≥75×10^9/L; Hemoglobin (Hb) ≥90 g/L (no blood transfusion within 14 days); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x upper limit of normal (ULN) (in patients with liver metastasis ≤5.0 x ULN); Total bilirubin ≤ 1.5 x ULN; Serum creatinine≤ 1.5 x ULN；
9. Male and female subjects of childbearing potential should agree to use suitable method of contraception during the treatment and 6 months after the last dose of study medication; female participants should have negative results of serum/urine pregnancy test within 7 days prior to enrollment and cannot be breastfeeding.

Exclusion Criteria:

1. Has participated in other clinical trials and received the treatment within 4 weeks prior to enrollment;
2. Patients who cannot swallow or have chronic diarrhea and intestinal obstruction, which may affect the administration and absorption of the drug;
3. Subject who meets one of the following criteria:

   * Corrected QT (QTc) ≥470ms in women, ≥450ms in men; or congenital long QT syndrome (LQTS), taking QT prolonging medications, and has a family history of long QT syndrome;
   * Resting ECG result shows clinically significant abnormalities of rhythm, conduction or morphology, requiring therapeutic intervention;
4. Urinalysis result shows protein in urine ≥ ++ and 24-hour urine protein > 1.0g;
5. Based on the investigator's assessment, patients with known severe comorbidities which may influence the safety of the patients and the study completion [such as uncontrolled hypertension (systolic pressure ≥150 mmHg or diastolic pressure ≥100 mmHg, despite treated with the optimal medicine), diabetes, etc.];
6. Patients who have symptoms of metastatic brain/meningeal tumors within 4 weeks of participation;
7. Ongoing adverse events>grade 1 at the time of participation (except hair loss and pigmentation);
8. Patients who have undergone major surgery or have not recovered from Invasive operation within 4 weeks prior to initiation of study treatment;
9. Coagulation disorders (INR >1.5, prothrombin time (PT) > ULN+4s or APTT >1.5ULN): with bleeding diathesis (such as active peptic ulcer) or receiving thrombolytic or anti-coagulant treatment;
10. Known pulmonary infection/ pneumonitis / interstitial pneumonia who are not suitable for the research;
11. Known active Hepatitis B or Hepatitis C virus infection;

    * if HBsAg result is positive, additional HBV DNA testing is required (the result is higher than the ULN of the research center);
    * if HCV antibody result is positive, additional HCV RNA testing is required (the result is higher than the ULN of the research center);
12. Known history of human immunodeficiency virus (HIV), or other acquired/congenital immune deficiency diseases or organ transplantation;
13. Other anti-tumor therapies are required (including radiotherapy, chemotherapy, immunotherapy, targeted treatment, traditional Chinese medicine, etc.);
14. Patients with known history of neurological or psychiatric disorders, including epilepsy or dementia;
15. Not suitable for the treatment assessed by the researchers;
16. Cardiac ejection fraction less than 50%;
17. Patients who have suffered from or are complicated with any other malignant tumor within 5 years (except radically resected skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, local prostate cancer, in situ cervical cancer or other carcinoma in situ).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of HA121-28 tablets in Advanced and/or Metastatic Cancer Refractory to Standard Treatment | At the end of Cycle 1 (each cycle is 28 days)
  MTD defined by dose limiting toxicities (DLTs) that occur in the first cycle. DLT defined as any clinically grade 3 or 4 non-hematologic toxicity as defined in the NCI CTC v4.0

SECONDARY OUTCOMES:
Antitumor Efficacy of HA121-28 tablets: RECIST criteria version 1.1. | up to 24 weeks
  Efficacy evaluation done using RECIST criteria version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Xu, Study Director — Clinical Medicine Department CSPC R&D Business Division
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Ruan DY, Huang WW, Li Y, Zhao Y, Shi Y, Jia Y, Cang S, Zhang W, Shi J, Chen J, Lin J, Liu Y, Xu J, Ouyang W, Fang J, Zhuang W, Liu C, Bu Q, Li M, Meng X, Sun M, Yang N, Dong X, Pan Y, Li X, Qu X, Zhang T, Yuan X, Hu S, Guo W, Li Y, Li S, Liu D, Song F, Tan L, Yu Y, Yu X, Zang A, Sun C, Zhang Q, Zou K, Dan M, Xu RH, Zhao H. Safety, pharmacokinetics and efficacy of HA121-28 in patients with advanced solid tumors and RET fusion-positive non-small-cell lung cancer: a multicenter, open-label, single-arm phase 1/2 trial. Signal Transduct Target Ther. 2025 Feb 28;10(1):62. doi: 10.1038/s41392-025-02155-5. PMID 40016191